CLINICAL TRIAL: NCT05367375
Title: Does Removing Patellofemoral Joint Osteophytes Reduce Anterior Knee Pain Following Unicompartment Knee Arthroplasty?
Brief Title: Comparison of Removing and Non-removing Patellofemoral Joint Osteophytes Following Medial Unicompartment Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Boonchana Pongcharoen, Associated professor, Thammasat University
Other Study IDs: MTU-EC-OT-0-224/62
Record Dates: First submitted 2022-05-01; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Anterior Knee Pain
Keywords: patellofemoral osteophyte; anteromedial osteoarthritis knee; mobile bearing UKA; patellofemoral pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- removing patellofemoral joint osteophytes: remove osteophyte at patella, medial femoral condyle and lateral femoral condyle
  Interventions: Procedure: removing osteophyte at patellofemoral joint
- non-removing patellofemoral joint osteophytes: no remove osteophyte at patella, medial femoral condyle and lateral femoral condyle

INTERVENTIONS:
Procedure: removing osteophyte at patellofemoral joint — to compare anterior knee pain between removing patellofemoral joint osteophytes and non-removing patellofemoral joint osteophytes after medial unicompartmental knee arthroplasty
  Groups: removing patellofemoral joint osteophytes

SUMMARY:
Background: Anterior knee pain (AKP) is a challenge following unicompartmental knee arthroplasty (UKA). Some surgeons remove patellofemoral joint (PFJ) osteophytes to reduce osteophyte impingement and AKP. However, there is evidence that PFJ osteophytes compensate for knee osteoarthritis (OA) by increasing and improving stability and increase contract surface area in knee osteoarthritis. Moreover, when PFJ osteophytes are not removed, some studies report good clinical outcomes. The issue of removing or leaving PFJ osteophytes is controversial.

The objective of this study was to compare AKP following mobile bearing UKA after removing or leaving PFJ osteophytes.

Methods: The prospective non-randomized study included 89 isolated medial osteoarthritis (OA) of knee. They were classified into 2 groups. Group (Gp)1 was removing PFJ osteophytes; consists of 44 knees. Gp2 was non-removing PFJ osteophytes: consists of 45 knees. The patients were follow up and recorded incidence of AKP and VAS for AKP at 6 weeks, 3months, 6 months, 1 year and 2 years. No patients were lost to follow up. The patellar tilt and shift were measured at 6 weeks, 3months, 6months, 1year and 2 years via skyline view radiography. The knee society scores, Oxford knee score, knee injury and osteoarthritis outcome score, forgotten joint score and Kujala scale also were recorede at 6 weeks, 3months, 6months, 1 year and 2 years.

DETAILED DESCRIPTION:
Removing and non-removing osteophyte at patellofemoral joint is controversial topic. The osteophyte may help to reduce load and improve stability of patellofemoral joint. Therefore, the purpose of this study is to compared anterior knee pain between removing and non-removing osteophyte at patellofemoral joint following medial mobile bearing unicompartmental knee arthroplasty

ELIGIBILITY:
Inclusion Criteria:

* age > 42 years old
* range of motion > 90 degrees
* flexion contracture< 15 degrees
* normal function of anterior cruciate ligament

Exclusion Criteria:

* spontaneous osteonecrosis of the knee
* inflammatory joinr arthritis
* full thickness cartilage loss at lateral compartment

Ages: 43 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: isolated medial osteoarthritis of the knee
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
incidence of anterior knee pain | 6 weeks
  number of participant that had anterior knee pain
incidence of anterior knee pain | 3 months
  number of participant that had anterior knee pain
incidence of anterior knee pain | 6 months
  number of participant that had anterior knee pain
incidence of anterior knee pain | 1 year
  number of participant that had anterior knee pain
incidence of anterior knee pain | 2 year
  number of participant that had anterior knee pain
Visual analogue scale for anterior knee pain | 6 weeks
  pain score 0= no pain and pain score 10= maximum pain
Visual analogue scale for anterior knee pain | 3 months
  pain score 0= no pain and pain score 10= maximum pain
Visual analogue scale for anterior knee pain | 6 months
  pain score 0= no pain and pain score 10= maximum pain
Visual analogue scale for anterior knee pain | 1 year
  pain score 0= no pain and pain score 10= maximum pain
Visual analogue scale for anterior knee pain | 2 years
  pain score 0= no pain and pain score 10= maximum pain

IPD SHARING:
Plan to Share IPD: No